CLINICAL TRIAL: NCT00001201
Title: Evaluation of Neuromuscular Diseases
Brief Title: Evaluation of Neuromuscular Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 840203; 84-N-0203
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-11

CONDITIONS: Healthy; Neuromuscular Disease; Peripheral Nervous System Disease
Keywords: Nerve Conduction Studies; EMG; Normal Volunteer; Electrophysiology; Peripheral Neuropathies; Myopathies
MeSH Terms: conditions — Neuromuscular Diseases; Peripheral Nervous System Diseases; Muscular Diseases

SUMMARY:
The peripheral nervous system is the portion of the nervous system outside of the brain and spinal cord. It includes the 12 pairs of cranial nerves, 31 pairs of spinal nerves and their branches, nerves responsible for sensation and maintenance of normal body functions (sympathetic and parasympathetic nerves).

Years of research using clinical examinations, microscopic examinations, and electrophysiology have made the peripheral nervous system the best-studied and most available portion of the nervous system. However, even with all of the extensive studies conducted on the peripheral nervous system, many conditions remain unclassified.

The EMG Laboratory at the NIH concentrates on studying disorders of the peripheral nervous system. This protocol was designed to allow the EMG Laboratory to;

I) Learn more about established diseases of the peripheral nervous system

II) Identify and characterize new diseases of the peripheral nervous system

III) Assess current techniques in the diagnosis of diseases of the peripheral nervous system

IV) Refine old methods and develop new ones for the diagnosis of diseases of the peripheral nervous system.

DETAILED DESCRIPTION:
Combined with careful clinical examination, electrophysiology and histopathology have rendered the peripheral nervous system the best studied and most accessible level of the nervous system. But even after intensive diagnostic evaluation of peripheral neuropathies in large diagnostic centers, 24 to 70% of disorders remain unclassified. Analogous statistics for disorders of muscle and neuromuscular transmission are not known but probably similar, if not worse. Clearly, detailed diagnostic characterization of disorders of the peripheral nervous system is the first stage in clinical intervention.

Currently, the EMG Laboratory at the NIH offers complete clinical, electrophysiologic, and, when appropriate, pathologic evaluations on all referrals from the other Branches and Institutes. Since these referrals come primarily from within the NIH, most disorders are secondary to other systemic disease. This protocol is designed to extend the services to direct referrals of primary disorders of the peripheral nervous system. The purposes are first, to learn more about established diseases; second, to identify and characterize new diseases; third, to assess current methodologies and technologies; and fourth, to refine old methods and develop new ones. Under this umbrella protocol, individual cases and clinical series can be investigated.

ELIGIBILITY:
Patients with disorders of the peripheral nervous system, including neuropathies, myopathies, or defective neuromuscular transmission.

Normal age-matched volunteers, including some from within a neurologic population.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500
Dates: Start 1984-10; Study Completion 2002-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Dyck PJ, Oviatt KF, Lambert EH. Intensive evaluation of referred unclassified neuropathies yields improved diagnosis. Ann Neurol. 1981 Sep;10(3):222-6. doi: 10.1002/ana.410100304. PMID 7294727
- [Background] Nielsen VK. Pathophysiology of hemifacial spasm: I. Ephaptic transmission and ectopic excitation. Neurology. 1984 Apr;34(4):418-26. doi: 10.1212/wnl.34.4.418. PMID 6322048
- [Background] Pollock M, Nukada H, Taylor P, Donaldson I, Carroll G. Comparison between fascicular and whole sural nerve biopsy. Ann Neurol. 1983 Jan;13(1):65-8. doi: 10.1002/ana.410130114. PMID 6830168